CLINICAL TRIAL: NCT02194881
Title: Ivacaftor in French Patients With Cystic Fibrosis and a G551D Mutation - Efficacy and Safety Results After the First Year of Treatment in the Real Life Setting.
Brief Title: Ivacaftor in French Patients With Cystic Fibrosis and a G551D Mutation
Acronym: IVACAFTOR1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: CCTIRS 13.652
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CFTR; G551D mutation; Novel treatments; Potentiator; Ivacaftor
MeSH Terms: conditions — Cystic Fibrosis | interventions — Therapeutics; ivacaftor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ivacaftor 1: patients with CF who are homozygous or heterozygous for the G551D mutation and treated with Ivacaftor
  Interventions: Drug: CF patients with a G551D mutation and treated with Ivacaftor

INTERVENTIONS:
Drug: CF patients with a G551D mutation and treated with Ivacaftor

SUMMARY:
The purpose of this study is to determine whether the treatment with Ivacaftor remains effective and safe in the patients with cystic fibrosis (and at least one G551D CFTR mutation) in the real life setting, after the drug has been approved by the Health authorities.

DETAILED DESCRIPTION:
The aims of our study are:

1. to describe the treated population at initiation of treatment,
2. to evaluate clinical parameters during the year before Ivacaftor was started, at initiation of treatment and during at least one year of treatment, until June 2014.
3. to evaluate the tolerance and safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* French patients with CF aged 6 or older who are homozygous or heterozygous for the G551D mutation
* Treated with Ivacaftor
* First prescription of Ivacaftor before June 1st 2013 (including patients randomized in the VX770 clinical trials)

Exclusion Criteria:

* CF patients younger than 6 years old
* CF patients who have received lung transplantation
* CF patients without a G551D mutation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CF aged 6 or older and cared in French CF centres
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
FEV1 (in liters and in % predicted) | until one years after initiation of treatment
  pulmonary function

SECONDARY OUTCOMES:
pulmonary exacerbations | until one years after initiation of treatment
number of hospitalizations and number of days of hospitalization per year | until one year after initiation of treatment
number of antibiotic treatments and number of days of antibiotic treatments | until one year after initiation of treatment
  number of oral antibiotic treatments and number of days of oral antibiotic treatments, number of IV courses and days of IV antibiotics per year
respiratory colonization | until least one year after initiation of treatment
  Evolution of bacteria and fungi in sputum
nutritional status | until one year after initiation of treatment
  Weight (and BMI-Zscore for children)
Adverse events | until one year after initiation of treatment
  Dates and reasons for interruption and discontinuation of treatment with Ivacaftor Adverse events, indicating what in the physician's opinion might be due to Ivacaftor

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hubert, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Result] Hubert D, Dehillotte C, Munck A, David V, Baek J, Mely L, Dominique S, Ramel S, Danner Boucher I, Lefeuvre S, Reynaud Q, Colomb-Jung V, Bakouboula P, Lemonnier L. Retrospective observational study of French patients with cystic fibrosis and a Gly551Asp-CFTR mutation after 1 and 2years of treatment with ivacaftor in a real-world setting. J Cyst Fibros. 2018 Jan;17(1):89-95. doi: 10.1016/j.jcf.2017.07.001. Epub 2017 Jul 12. PMID 28711222